CLINICAL TRIAL: NCT02539342
Title: Caphosol Study: A Randomized Controlled Open-Labeled Trial Investigating Topical Caphosol for Prevention of Oral Mucositis in Children, Adolescents and Young Adults Receiving Chemotherapy
Brief Title: Caphosol Study: Prevention of Oral Mucositis in Children, Adolescents and Young Adults Receiving Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Burke, Associate Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Caphosol Study
Record Dates: First submitted 2015-08-20; First posted 2015-09-03 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Cancer; Chemotherapy
MeSH Terms: conditions — Stomatitis; Neoplasms | interventions — Saliva, Artificial; Biotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caphosol Arm (Experimental): Caphosol Arm: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day from the start of chemotherapy until 7 days after the completion of chemotherapy AND until the ANC is >500 after count recovery OR until the the symptoms or oral mucositis resolve, whichever occurs last. Patients will also complete a study diary to record symptoms of oral mucositis.
  Interventions: Drug: Caphosol
- Control Arm (Active Comparator): Control Arm: Subjects randomized to the Control Arm will use Biotene 4 times per day. They will also complete a study diary to record doses and any symptoms of oral mucositis. This will begin at the start of chemotherapy until for 7 days AND until ANC >500 after nadir or oral mucositis resolves (whichever occurs later)
  Interventions: Drug: Biotene

INTERVENTIONS:
Drug: Caphosol — Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day as follows:
  * Each dose consists of two 15 mL syringes, to be mixed at time of administration. Caphosol must be used within 15 minutes of mixing.
    o Participants may increase the use to 6 times per day if you have symptoms of mucositis.
  * Using one of the syringes, rinse and gargle (if patient is able) for one minute and then spit. Repeat using the remaining syringe.
    * For younger patients (less than or equal to 6 years of age), volume may be reduced to two syringes containing 5-10 mL each.
    * For patients unable to successfully rinse and spit, caregivers may paint their mouth (using medical sponge swabs) with the solution two times. Repeat using the second syringe.
  * Patients are to avoid other oral medications, other mouth cares and food or drink for 15 minutes after using Caphosol.
  * Patients may use Biotene (5-10 mL) to swish and spit after the 15 minutes has passed
  Other Names: artificial saliva; Supersaturated calcium phosphate rinse
  Arms: Caphosol Arm
Drug: Biotene — • Use 5 to 10 mL of Biotene to swish and spit
  o For patients unable to successfully rinse and spit, caregivers may paint their mouth (using medical sponge swabs) with the solution two times. Prior to swabbing the patient's mouth, pour Biotene into a cup and using the medical sponge, soak up the solution and use the swab to coat the inside of the patient's mouth. Repeat with a second swab.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to determine if the administration of Caphosol rinse, at the start of chemotherapy, will prevent the development of mucositis (greater than or equal to grade 2 in children, adolescents and young adults. This is a randomized, controlled trial.

DETAILED DESCRIPTION:
Oral mucositis, is a common and debilitating complication of cancer therapy. It is an inflammatory injury to the epithelial and sub-epithelial cells of the oral mucosa. The incidence and severity of oral mucositis depends on many factors including the age and diagnosis of the patient, the specific treatment regimen, underlying oral hygiene and genetic factors 2-4. This ranges from around 40% of patients getting chemotherapy for solid tumors to 70-90% of patients getting chemotherapy for before stem cell transplant.

Oral mucositis causes significant pain, interferes with eating, talking and swallowing, significantly diminishes enteral nutritional intake and has a substantial negative impact on quality of life. Patients may require hospitalization for management of the complications of mucositis, including poor nutrition, dehydration and pain. Injury to the oral mucosa also increases the risk of systemic infections. Finally, the development of oral mucositis may require delays or dose reductions in future chemotherapy courses, potentially jeopardizing disease cure rates.

Despite all that is known about the mechanism, course and complications of oral mucositis, there are no consensus guidelines on prevention or treatment of chemotherapy-induced oral mucositis and there is significant variation on approach to mucositis across treatment centers.

Caphosol (Jazz Pharmaceuticals, Inc. Palo Alto, CA) was designed in part to replace the normal ionic and pH balance of the oral cavity and been used to prevent and/or treat oral mucositis. Caphosol is hypothesized to diffuse into epithelial intracellular spaces and permeate mucosal lesions in oral mucositis.

This study is a randomized, controlled trial evaluating the use of topical Caphosol therapy to prevent oral mucositis (Grade ≥ 2) in children, adolescents and young adults undergoing chemotherapy. At the time of enrollment, patients will be randomized to either the control arm or the Caphosol arm. The treatment period will extend from the start of chemotherapy and continue for 7 days after completion of chemotherapy AND until the ANC is > 500 after nadir (count recovery) or until the symptoms of oral mucositis resolve; whichever occurs last.

Study patients will be recruited from the MACC Fund Center and the oncology inpatient service. Study entry is open to patients regardless of gender or ethnic background. While there will be every effort to seek out and include females and minority patients, the patient population is expected to be no different than that of other oncology studies at the Medical College of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Oncology patients, at initiation of their oncology therapy, who are at risk of developing oral mucositis during their scheduled cancer therapy, defined by meeting one or more of the following criteria:
* Patients receiving one or more of the following chemotherapy agents:

  * Actinomycin D
  * Carboplatin
  * Cisplatin
  * Cytarabine at doses > 1 gram/m2
  * Daunorubicin
  * Doxorubicin
  * Methotrexate at doses > 1 gram/m2
  * Mitoxantrone
* Age 0 to 25 years
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Patients receiving glutamine treatment for oral mucositis.
* Patients undergoing autologous or allogeneic hematopoietic cell transplantation are excluded from this study.
* Patients receiving concurrent Head & Neck radiation therapy or within 6 weeks of completion of radiation therapy.
* Pregnant or lactating patients. The agent used in this study is not known to be teratogenic to a fetus, but has not been studies, and there is no information on the excretion of the agent into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Known allergy to Caphosol

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Burke, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caphosol Arm: Caphosol Arm: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day from the start of chemotherapy until 7 days after the completion of chemotherapy AND until the ANC is >500 after count recovery OR until the the symptoms or oral mucositis resolve, whichever occurs last. Patients will also complete a diary to record symptoms of oral mucositis.
  Caphosol: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day as follows:
  * Each dose consists of two 15 mL syringes, to be mixed at time of administration. Caphosol must be used within 15 minutes of mixing.
    o Participants may increase the use to 6 times per day if you have symptoms of mucositis.
  * Using one of the syringes, rinse and gargle (if patient is able) for one minute and then spit. Repeat using the remaining syringe.
    * For younger patients (less than or equal to 6 years of age), volume may be reduced to two syringes containing 5-10 mL each.
    * For patients unable to successfu
- Control Arm: Control Arm: Subjects randomized to the Control Arm will use Biotene 4 times per day. They will also complete a study diary to record doses and any symptoms of oral mucositis. This will begin at the start of chemotherapy until for 7 days AND until ANC >500 after nadir or oral mucositis resolves (whichever occurs later)
  Biotene: • Use 5 to 10 mL of Biotene to swish and spit
  o For patients unable to successfully rinse and spit, caregivers may paint their mouth (using medical sponge swabs) with the solution two times. Prior to swabbing the patient's mouth, pour Biotene into a cup and using the medical sponge, soak up the solution and use the swab to coat the inside of the patient's mouth. Repeat with a second swab.
Period: Overall Study
Arm/Group | Caphosol Arm | Control Arm
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We had only 1 enrollment overall and that was to the Caphosol arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Caphosol Arm | Control Arm | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure the Development of Oral Mucositis (Grade >/= 2) in Children, Adolescents and Young Adults.
Description: The development of Mucositis Grade >/= 2 in children receiving chemotherapy as evaluated using CTCAE 4.0
Time Frame: 24 months
Population: We only had 1 patient enrolled on the Caphosol Arm and none on the Control Arm
Measure: Count of Participants; unit: Participants
Groups:
- Caphosol Arm: Caphosol Arm: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day from the start of chemotherapy until 7 days after the completion of chemotherapy AND until the ANC is >500 after count recovery OR until the the symptoms or oral mucositis resolve, whichever occurs last. Patients will also complete a study diary to record symptoms of oral mucositis.
  Caphosol: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day as follows:
  * Each dose consists of two 15 mL syringes, to be mixed at time of administration. Caphosol must be used within 15 minutes of mixing.
  * Using one of the syringes, rinse and gargle (if patient is able) for one minute and then spit. Repeat using the remaining syringe.
  * Patients may use Biotene (5-10 mL) to swish and spit after the 15 minutes has passed
Arm/Group | Caphosol Arm | Control Arm
Number analyzed (Participants) | 1 | 0
Participants
  Mucositis Grade >/= 2 | 1 | 0
  Mucositis Grade </=2 | 0 |

2. Other Pre Specified Outcome: Tolerability of Four Times Daily Caphosol Therapy
Description: Any adverse events attributable to caphosol therapy being given 4 times daily
Time Frame: 24 months
Population: 1 patient enrolled on Caphosol and None on Control Arm
Measure: Number; unit: events
Arm/Group | Caphosol Arm | Control Arm
Number analyzed (Participants) | 1 | 0
events | 0 |

ADVERSE EVENTS:
Time Frame: 4 months - but there were no adverse events
Description: There were no adverse events
Groups:
- Caphosol Arm: Caphosol Arm: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day from the start of chemotherapy until 7 days after the completion of chemotherapy AND until the ANC is >500 after count recovery OR until the the symptoms or oral mucositis resolve, whichever occurs last. Patients will also complete a study diary to record symptoms of oral mucositis.
  Caphosol: Subjects randomized to the Caphosol Arm will use Caphosol 4 times per day as follows:
  • Each dose consists of two 15 mL syringes, to be mixed at time of administration. Caphosol must be used within 15 minutes of mixing.
  o
  • Patients may use Biotene (5-10 mL) to swish and spit after the 15 minutes has passed
Arm/Group | Caphosol Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02539342/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02539342/ICF_001.pdf